CLINICAL TRIAL: NCT05797350
Title: Paul Glaucoma Implant Versus Ahmed Glaucoma Valve in Childhood Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Watany Eye Hospital (Other)
Collaborators: Moorfields Eye Hospital Centre Abu Dhabi (Other)
Responsible Party: Principal Investigator, Mohamed El Baharwy, Clinical Professor, Al Watany Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlWatanyEyeH
Record Dates: First submitted 2023-03-12; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paul Glaucoma Implant (Active Comparator): The Paul glaucoma implant (PGI) will be used as an active comparator group to compare its effectiveness and safety with the Ahmed glaucoma valve in the treatment of childhood glaucoma. The PGI works by diverting excess fluid from the eye to a plate placed under the conjunctiva, which allows the fluid to drain away from the eye and be absorbed. This helps to lower the pressure inside the eye, which is important for preventing vision loss and other complications associated with glaucoma.
  The PGI has a smaller internal and external tube diameter than the Ahmed glaucoma valve, which reduces the contact area between the tube and the corneal endothelium. This theoretically reduces the rate of endothelial cell loss, which can be a complication of GDDs. Additionally, the extraocular portion of the PGI is smaller, which may reduce the long-term risk of tube erosion and exposure.
  The smaller lumen may theoretically reduce the risk of postoperative hypotony as well.
  Interventions: Device: Glaucoma Drainage Device
- Ahmed Glaucoma valve (Active Comparator): The Ahmed glaucoma valve (AGV) arm of the study is the active comparator group and is intended to be directly compared to the Paul glaucoma implant (PGI) in treating childhood glaucoma. The AGV is a type of glaucoma drainage device that is designed to lower intraocular pressure in patients with refractory glaucoma. It is made of a rigid plastic material and consists of a small drainage tube that is inserted into the eye and a valve mechanism that helps regulate the flow of aqueous humor from the eye to the external drainage tube.
  The AGV is implanted during a surgical procedure, and its design allows it to be placed in a variety of locations in the eye. The valve mechanism helps to regulate the flow of aqueous humor, and the device is designed to be long-lasting with a low risk of complications. The AGV is a well-established treatment option for patients with refractory glaucoma and has been used for many years in clinical practice.
  Interventions: Device: Glaucoma Drainage Device

INTERVENTIONS:
Device: Glaucoma Drainage Device — Both the Paul glaucoma implant (PGI) and Ahmed glaucoma valve (AGV) are types of glaucoma drainage devices (GDDs) used to lower intraocular pressure in patients with refractory glaucoma. Devices will be implanted during a surgical procedure and work by diverting excess fluid from the eye to an external drainage tube, allowing the fluid to drain away from the eye and be absorbed into the surrounding tissue. This will help to lower the pressure inside the eye, which is important for preventing vision loss and other complications associated with glaucoma.

SUMMARY:
A randomized controlled trial comparing the efficacy and safety of Paul glaucoma implant and Ahmed glaucoma valve in refractory childhood glaucoma patients

DETAILED DESCRIPTION:
A prospective randomized controlled trial was conducted at Al Watany Eye Hospital in Egypt. Patients with refractory primary or secondary childhood glaucoma who glaucoma specialist has decided to perform a tube implant to control their intraocular pressure are randomized to receive either Paul or Ahmed glaucoma drainage devices.

Patients will be followed up for at least one year during which the following data are collected.

Age, sex, laterality, preoperative and postoperative intraocular pressure and glaucoma medications at 1,3,6, 9, and 12 months visits. Any intraoperative or postoperative complications will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Childhood glaucoma patients (whether primary or secondary) including Juvenile open angle glaucoma if the age at the time of surgery was ≤18 years.
* The included patients are those with refractory glaucoma who require a tube to control their intraocular pressure.

Exclusion Criteria:

* Any patient with incomplete data or has a follow-up less than 1 year will be excluded from the study.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
IOP Reduction | 1 year
  More than 20% change from baseline without development of vision threatening complications

SECONDARY OUTCOMES:
Glaucoma Medication Alterations | 1 year
  Assessment of changes in number of medications for IOP reduction after procedure (i.e., did patients have a reduction or gain in use of medications to reduce their IOP after the procedure?)
Post-operative complications | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Maadi eye subspeciality center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No